CLINICAL TRIAL: NCT00333424
Title: A Randomised, Placebo-Controlled, Double-Blind, Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of a Candidate Prophylactic pHIS-HIV-AE DNA Prime and rFPV-HIV-AE Boost HIV Vaccination Strategy
Brief Title: Thai Prophylactic HIV Vaccine Phase I Study
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Vaccines safe but not immunogenic in 8 participants; trial closed to further recruitment by the protocol steering committee & DSMB.
Sponsor: Kirby Institute (Other Government)
Collaborators: Thai Red Cross AIDS Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NCHECR-AE1; NCT00476749 (obsolete NCT alias); NCT00859248 (obsolete NCT alias); NCT00859820 (obsolete NCT alias)
Record Dates: First submitted 2006-06-01; First posted 2006-06-05 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: HIV
Keywords: HIV; Human Immunodeficiency Virus; Prophylactic vaccine
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Vaccines, DNA; PRIME protocol; Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Placebo (Placebo Comparator): placebo containing diluent alone
  Interventions: Biological: pHIS-HIV-AE (DNA vaccine) prime and rFPV-HIV-AE (recombinant fowlpox virus boost) vaccine

INTERVENTIONS:
Biological: pHIS-HIV-AE (DNA vaccine) prime and rFPV-HIV-AE (recombinant fowlpox virus boost) vaccine — 6mg pHIS-HIV-AE at weeks 0, 4 and 8; 3 x 10e8 pfu/mL rFPV-HIV-AE at week 12

SUMMARY:
The development of a safe and effective vaccine for HIV is the subject of intensive world-wide research. Various approaches are being investigated in monkey models and humans. This is a randomized, double-blind trial to evaluate the safety and immunogenicity of a candidate preventative human immunodeficiency virus (HIV) vaccine strategy in 24 healthy adult Thai volunteers with no identifiable risk behaviour for HIV-1 infection. Volunteers will receive three "priming" vaccinations at weeks 0, 4 and 8 (pHIS-HIV-AE, a DNA vector delivering AE clade HIV-1 genes). This will be followed at week 12 by single "boost" vaccination (rFPV-HIV-AE, non-replicating, recombinant fowlpox virus vector delivering the same HIV-1 genes). Safety and immunological monitoring will continue to 52 weeks

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, as judged by the screening physician based on medical history, physical examination and laboratory results
* 18 - 55 years of age, inclusive
* Laboratory blood values within clinically acceptable range
* Women of reproductive potential must have a negative urine beta-human chorionic gonadotropin (B-HCG) pregnancy test at both the screening and baseline visits
* Agreement to employ barrier contraception for 4 weeks preceding entry and for the whole duration of the study (52 weeks)
* Agreement to undertake HIV testing and to receive results
* Provision of written informed consent approved by the Institutional Ethics Committee (IEC).

Exclusion Criteria:

* HIV positive
* HBsAg or HCV positive
* Identifiable risk behaviour for HIV infection, defined as any one of the following:

  * sexual partners of HIV positive people
  * individuals reporting unprotected intercourse with a partner of unknown HIV status, if that partner is reported to be at higher risk for HIV infection ("higher risk of HIV infection" is defined as individuals reporting unprotected anal intercourse (UAI), unprotected intercourse with sex workers and/or sharing injecting equipment within the 12 months preceding trial entry
  * men reporting any UAI with male partners of unknown status in the 12 months preceding entry to the study
  * individuals who in the 12 months preceding entry to the study have been diagnosed with a new sexually transmissible infection (STI) that may have been acquired through anal or vaginal intercourse (receptive or insertive)
  * individuals reporting sharing of injecting equipment in the last 12 months
* Recipients of prior HIV candidate vaccines in a previous HIV vaccine trial (does not apply to volunteers who received placebo or adjuvant in such a trial)
* Recipients of live attenuated vaccines within 60 days prior to entering the study. Whole killed, toxoid or sub-unit vaccines e.g. influenza, pneumococcus, tetanus, hepatitis B are not exclusionary when given at least 4 weeks prior to the scheduled experimental HIV vaccines
* Known or suspected hypersensitivity to egg products or a known history of anaphylaxis or any other serious adverse reactions to any vaccinations
* History of serious allergic reactions requiring hospitalisation or emergency medical care (e.g. Steven-Johnson's syndrome, bronchospasm or hypotension) to any substance
* Clinically significant intercurrent illness or a history of clinically significant illness requiring immunomodulatory (including corticosteroids) or cytotoxic treatment (e.g. cancer) or any significant disease conditions that in the opinion of the Principal Investigator precludes the individual from participating in the study
* Recipients of blood products or immunoglobulins within 6 months prior to entering the study
* Recipients of experimental or investigational agents within 30 days prior to entering the study
* Recreational and/or therapeutic drug-use that, in the opinion of the Principal Investigator, might compromise the volunteer's participation in any way
* Medical or psychiatric condition or occupational responsibilities that may preclude compliance with the protocol
* Pregnant or lactating women, or women planning to become pregnant during the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
All safety data summarised & compared by randomly assigned vaccination group. Primary immunological outcome is mean difference in change in percent of IFN-y + CD4+ and/or CD8+ cells by intracellular cytokine staining (ICCS) from week 0 to 13. | 13 weeks

SECONDARY OUTCOMES:
Proportion of patients with positive ICCS assay responses; peripheral blood mononuclear cell responses to HIV antigens; proportion of patients with positive ELIspot assay responses; anti-HIV Gag, Pol & Env antibodies. | week 13

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD PhD, Principal Investigator — HIV-NAT, Thai Red Cross AIDS Research Center
Locations (1):
- HIV-NAT (The HIV Netherlands Australia Thailand Research Collaboration), Thai Red Cross AIDS Research Centre, Bangkok, Thailand

REFERENCES:
- [Result] Hemachandra A, Puls RL, Sirivichayakul S, Kerr S, Thantiworasit P, Ubolyam S, Cooper DA, Emery S, Phanuphak P, Kelleher A, Ruxrungtham K. An HIV-1 clade A/E DNA prime, recombinant fowlpox virus boost vaccine is safe, but non-immunogenic in a randomized phase I/IIa trial in Thai volunteers at low risk of HIV infection. Hum Vaccin. 2010 Oct;6(10):835-40. doi: 10.4161/hv.6.10.12635. Epub 2010 Oct 1. PMID 20864808